CLINICAL TRIAL: NCT05874999
Title: Feasibility and Acute Effects of Supramaximal High-Intensity Interval Training in People With COPD
Brief Title: Acute Effects of Supramaximal High-Intensity Interval Training in People With COPD
Acronym: COPD-HIIT-AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Heart Lung Foundation (Other); Riksförbundet HjärtLung (Unknown)
Responsible Party: Principal Investigator, Andre Nyberg, Associate Professor, Umeå University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: COPD-HIIT ACUTE
Record Dates: First submitted 2023-03-30; First posted 2023-05-25 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: COPD; Healthy Older Adults
Keywords: Acute Exercise; High-intensity Interval Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Obstructive Pulmonary Disease (COPD) (Experimental): People with chronic obstructive pulmonary disease (COPD) (n = 16)
  Interventions: Other: Supramaximal High-Intensity Interval Training at 60% of MPO6; Other: Moderate-Intensity Continuous Training; Other: Supramaximal High-Intensity Interval Training at 80% of MPO6
- Healthy Controls (HC) (Active Comparator): Healthy controls matched on age, sex and objectively measured physical activity (n = 16)
  Interventions: Other: Supramaximal High-Intensity Interval Training at 60% of MPO6; Other: Moderate-Intensity Continuous Training; Other: Supramaximal High-Intensity Interval Training at 80% of MPO6

INTERVENTIONS:
Other: Supramaximal High-Intensity Interval Training at 60% of MPO6 — Supramaximal HIIT is performed as 10×6 second intervals against a load of 60% of maximum mean power output for 6 seconds (MPO6) with a 54 second recovery between intervals. The MPO6 was estimated from the BCST.
  Duration supramaximal HIIT: 10 minutes
  Warm-up and cool-down: 5 minutes at 30% of maximum aerobic power (MAP) obtained during maximal incremental cardiopulmonary exercise test (CPET) on a stationary bicycle.
  Other Names: Supramaximal High-Intensity Interval Training at 60% of MPO6 (HIIT60%)
Other: Moderate-Intensity Continuous Training — MICT is performed against a load of 60% of MAP obtained during a maximal incremental CPET on a stationary bicycle.
  Duration MICT: 20 minutes
  Warm-up and cool-down: 5 minutes at 30% of MAP obtained during maximal incremental CPET on a stationary bicycle.
  Other Names: MICT
Other: Supramaximal High-Intensity Interval Training at 80% of MPO6 — Supramaximal HIIT is performed as 10×6 second intervals against a load of 80% of MPO6 with a 54 second recovery between intervals. The MPO6 was estimated from the BCST.
  Duration supramaximal HIIT: 10 minutes
  Warm-up and cool-down: 5 minutes at 30% of MAP obtained during maximal incremental CPET on a stationary bicycle.
  Other Names: Supramaximal High-Intensity Interval Training at 80% of MPO6 (HIIT80%)

SUMMARY:
High-intensity exercise is essential for optimal development of cardiorespiratory fitness and health. This is, however, challenging for most people with chronic obstructive pulmonary disease (COPD) due to ventilatory limitations, leading to exercise at lower intensities accompanied by suboptimal stress on the cardiovascular and muscular system.

The aims of this cross-over trial is:

1. To compare the acute effects of short-duration supramaximal high-intensity interval training (HIIT) vs. traditional moderate-intensity continuous training (MICT) in people with COPD and matched healthy controls (HC).
2. To investigate the feasibility of supramaximal HIIT in people with COPD and matched HC.
3. To compare the cardiorespiratory demand, exercise intensity and symptoms during a modified Borg Cycle Strength Test (BCST) and a cardiopulmonary exercise test (CPET) in people with COPD and HC.

DETAILED DESCRIPTION:
In this study, eligible participants attended the facility four times within 14 days with at least 48 hours of rest between visits.

Exercise tests (visit 1, week 1):

After pulmonary functions tests, a CPET on a stationary bicycle was performed according to international guidelines. After 1.5 hours of recovery, a BCST was performed to assess anaerobic exercise capacity and determine exercise intensities for supramaximal HIIT.

Exercise sessions (visit 2 - week 1; visit 3 - week 2; visit 4 - week 2):

The order of the two first exercise sessions (HIIT at 60% of MPO6 or MICT) on a stationary bicycle were randomized. The exercise session at HIIT at 80% of MPO6 was always the third exercise session.

During all exercise sessions, blood collection was performed at baseline after a 15-minute seated rest. During HIIT, blood was collected immediately after, and 30 minutes after the 10-minute HIIT period. For MICT, blood was collected after 10 minutes (isotime in relation to HIIT), immediately after, and 30 minutes of cycling at 60% MAP.

ELIGIBILITY:
COPD

Inclusion Criteria:

* COPD with non-reversible airflow obstruction diagnosis (post-bronchodilator forced expiratory volume during the first second/forced vital capacity (FEV1/FVC) < 0.7)
* Age: > 40 years

Exclusion Criteria:

* Recent exacerbation of COPD (< 6 weeks)
* Neuromuscular, orthopaedic and/or any other condition that can compromise participation in testing
* Recent lung cancer (< 5 years)
* Unstable cardiac disease and/or cardiac stimulator

HC

Inclusion Criteria:

- Age: > 40 years

Exclusion Criteria:

* Neuromuscular, orthopaedic and/or any other condition that can compromise participation in testing
* Any respiratory disease
* Recent lung cancer (< 5 years)
* Unstable cardiac disease and/or cardiac stimulator
* Too low or high physical activity level that prohibits matching

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Exercise intensity | During visit 2 (week 1)
  Produced watt at the set training intensity
Exercise intensity | During visit 3 (week 2)
  Produced watt at the set training intensity
Exercise intensity | During visit 4 (week 2)
  Produced watt at the set training intensity
Brain-derived neurotrophic factor (BDNF) | During visit 2 (week 1)
  Concentration of BDNF in obtained venous blood samples before, during and after exercise. Measured as ng/mL or pg/mL.
Brain-derived neurotrophic factor (BDNF) | During visit 3 (week 2)
  Concentration of BDNF in obtained venous blood samples before, during and after exercise. Measured as ng/mL or pg/mL.
Brain-derived neurotrophic factor (BDNF) | During visit 4 (week 2)
  Concentration of BDNF in obtained venous blood samples before, during and after exercise. Measured as ng/mL or pg/mL.

SECONDARY OUTCOMES:
Cardiorespiratory demand | During visit 1 (CPET and BCST; week 1), visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Gas exchange parameters (e.g. VO2, VCO2, ventilatory equivalents, RER) and lung volumes (e.g. VE, Vt, breathing frequency) obtained with a metabolic cart (breath by breath methodology) and heart rate (beats per minutes) during exercise during exercise.
Venous blood lactate concentration | During visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Measured before, during and after exercise.
Rating of perceived exertion | During visit 1 (CPET and BCST; week 1), visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Rating of perceived exertion scale (Borg RPE). Minimum value = 6 Maximum value = 20 A higher score means higher exertion.
Rating of symptoms | During visit 1 (CPET and BCST; week 1), visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Rating of dyspnea and leg fatigue symptoms via Borg CR (category ratio) 10 during exercise Minimum value = 0 Maximum value = 10 A higher score means higher severity of symptoms
Peripheral blood oxygen saturation (SpO2) | During visit 1 (CPET and BCST; week 1), visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  SpO2 during exercise
Blood pressure | During visit 1 (CPET and BCST; week 1), visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Systolic and diastolic blood pressure during exercise
Circulating levels of neurotrophic factors | During visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Plasma or serum concentration (measured as mg/l, ng/l, or pq/l) of irisin, cathepsin B, clusterin, in obtained venous blood samples before, during and after exercise.
Circulating levels of exerkines | During visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Plasma or serum concentration of interleukin (IL)-1b, IL-4, IL-6, IL-8, IL-10, IL-13, IL-15, IL-17, tumor necrosis factor (TNF)-α, vascular endothelial growth factor (VEGF), hepatocyte growth factor (HGF), and adiponectin in obtained venous blood samples before, during and after exercise.
Exercise session completion | During visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Number of uninterrupted exercise sessions
Exercise preference | At the end of visit 3 (week 2)
  Preference for HIIT at 60% of MPO6 or MICT, defined as answer on the following question:
  "If the MICT and HIIT would be equally effective in improving your health and physical capacity, which one would you prefer to perform?"
Session RPE | During visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Rating of session RPE on Borg CR (category ratio) 10 is assessed 30 min after every exercise session Minimum value = 0 Maximum value = 10 A higher score means higher session exertion
Exercise capacity | During visit 1 (CPET; week 1)
  Maximal aerobic power (MAP) expressed as produced watt at VO2peak
Exercise intensity | During visit 1 (BCST; week 1)
  Maximum mean power output for 30 seconds (MPO30) in watts
Adverse events | During visit 2 (week 1), visit 3 (week 2) and visit 4 (week 2)
  Occurence and severity of adverse events. The severity of adverse events will be assessed and rated into four different categories: 1) minor and temporary, 2) serious symptoms (potential risk of severe injury or life threatening, 3) manifest injury or disease and 4) death. An adverse event rate will be calculated for each participant as the total number of sessions during which any adverse events occurred divided by the total number of attended sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Nyberg, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if individual participant data (IPD) will be available to other researchers.